CLINICAL TRIAL: NCT04526184
Title: Systemic Effects of A Continuous Blood Flow Restricted Aerobic Exercise Session in COPD Patients: A Randomised Controlled Trial.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ahmet Gunes, PhD Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMU
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups will be formed as healthy and patient groups and the same treatment initiative will be applied.
Who Masked: Participant, Outcomes Assessor
Masking Description: 25 COPD patients were referred to the study from the pulmonology clinic of the hospital where the study was conducted by a medical secretary who was blinded to the intervention. In addition, 21 healthy individuals volunteered to participate in the study from the same hospital where the study was previously announced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy group (Active Comparator): 25 healthy individuals between the ages of 40-70 will be contacted by phone and included in the initiative.
  Interventions: Procedure: aerobic exercise with blood flow restriction
- patient group (Active Comparator): 25 individuals will be selected randomly from 103 patients with COPD from hospital records.
  Interventions: Procedure: aerobic exercise with blood flow restriction

INTERVENTIONS:
Procedure: aerobic exercise with blood flow restriction — Patients and healthy individuals will be given 30 minutes of aerobic exercise by cycling, by restricting lower extremity blood flow.

SUMMARY:
Patients with COPD that a pulmonologist classifies between Stage 1-2 in accordance with the GOLD criteria and age and gender-matched healthy individuals will be included in the study.

In both groups (n = COPD: 17, Healthy: 17), aerobic exercise (AE) in the target heart rate range of 50% intensity, performed by cycling accompanied by blood flow restriction, will be applied.

DETAILED DESCRIPTION:
Target heart rate will be calculated from the formula "(Maximal heart rate-resting heart rate) x% desired intensity ratio + resting heart rate".

The target occlusion amount in the lower extremity will be calculated by calculating 45% of the complete occlusion rates reported by Michael et al. The proximal border of the thigh cuffs will be tied in line with the gluteal lines on both sides.

Exercise tolerance and dyspnea condition; Measurement properties in COPD will be evaluated using a well-defined modified Borg scale (MBS). Individuals will use any bronchodilator that their doctor sees fit before trying.

The target aerobic exercise intensity will be reached in the last minute of the first five-minute warm-up period by maintaining a 4-6 feeling of dyspnea in the MBS, by increasing pedal resistance and speed. In case of extreme shortness of breath, exercise intensity will be reduced to resting heart rate.

In the event of oxygen desaturation (85%) during the intervention, the intervention will be terminated.

Aerobic exercise training protocol; It was planned as 50 rpm speed and warming up at the lowest pedal resistance during the first 4 minutes, reaching the target exercise intensity range in the next 1 minute, aerobic training at the target heart rate range and appropriate MBS value for the next 20 minutes, cooling down in the last 5 minutes. The duration will be reduced in case of excessive shortness of breath, fatigue and muscle pain due to increased exercise volume. The distance, calories, and maximum speed values measured during the study will be recorded.

Before and immediately after the study, all participants had muscle damage (creatine kinase), anti-inflammatory response (CRP, neutrophil), oxidative stress response (uric acid, LDH), oxygen saturation, heart rate, systolic and diastolic pressure will be examined.

Institution of the Study: Karabuk University Research Hospital Chest Diseases Clinic Center / Karabuk. The study would be conducted in the presence of a chest diseases specialist.

ELIGIBILITY:
Inclusion Criteria:

* No drug change for at least 30 days for the COPD group
* Not participating in a structured activity program for at least six months
* Have the ability to cooperate

Exclusion Criteria:

* Presence of any pathology that limits physical activity performance
* Presence of severe or unstable heart disease
* Presence of peripheral artery disease
* Being in an exacerbation period of the disease
* Presence of another active disease (rheumatic, oncological, traumatic etc.)
* Any neurological or orthopedic disease that prevents exercise

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Because COPD is generally more common in males, patients of this gender were included in the study.
Enrollment: 46 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-03-19 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
creatine kinase | 30 minutes
  rhabdomyolysis marker
C reactive protein, neutrophil | 30 minutes
  inflammatory marker
oxygen saturation | 30 minutes
  blood oxygen saturation
heart rate | 30 minutes
  determination of aerobic exercise dose
systolic and diastolic pressure | up to 18 weeks
  to mean arterial pressure calculation
modified borg scale | up to 18 weeks.
  dyspnoea measurement, Minimum 1, maximum 7 points are obtained. 5 indicates the best respiratory condition, 10 the worst respiratory condition.
oxidative stress markers | up to 18 weeks
  uric acid, lactate dehydrogenase

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük Üniversitesi Araştırma Hastanesi Göğüs Hastalıkları Kliniği, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Result] Kacin A, Strazar K. Frequent low-load ischemic resistance exercise to failure enhances muscle oxygen delivery and endurance capacity. Scand J Med Sci Sports. 2011 Dec;21(6):e231-41. doi: 10.1111/j.1600-0838.2010.01260.x. Epub 2011 Mar 8. PMID 21385216
- [Result] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Result] Nolan CM, Rochester CL. Exercise Training Modalities for People with Chronic Obstructive Pulmonary Disease. COPD. 2019 Dec;16(5-6):378-389. doi: 10.1080/15412555.2019.1637834. Epub 2019 Nov 4. PMID 31684769
- [Result] Loenneke JP, Allen KM, Mouser JG, Thiebaud RS, Kim D, Abe T, Bemben MG. Blood flow restriction in the upper and lower limbs is predicted by limb circumference and systolic blood pressure. Eur J Appl Physiol. 2015 Feb;115(2):397-405. doi: 10.1007/s00421-014-3030-7. Epub 2014 Oct 22. PMID 25338316
- [Result] Wilson JM, Lowery RP, Joy JM, Loenneke JP, Naimo MA. Practical blood flow restriction training increases acute determinants of hypertrophy without increasing indices of muscle damage. J Strength Cond Res. 2013 Nov;27(11):3068-75. doi: 10.1519/JSC.0b013e31828a1ffa. PMID 23446173
- [Result] Berzosa C, Cebrian I, Fuentes-Broto L, Gomez-Trullen E, Piedrafita E, Martinez-Ballarin E, Lopez-Pingarron L, Reiter RJ, Garcia JJ. Acute exercise increases plasma total antioxidant status and antioxidant enzyme activities in untrained men. J Biomed Biotechnol. 2011;2011:540458. doi: 10.1155/2011/540458. Epub 2011 Mar 9. PMID 21436993